CLINICAL TRIAL: NCT00183612
Title: Developmental Pharmacokinetics of Psychotropic Drugs: Olanzapine
Brief Title: Determining the Safety and Effectiveness of Olanzapine in Children and Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Maurizio Fava, MD, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K08MH001765 (NIH); K08MH001765 (NIH); DSIR CT-M
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar Disorder; Psychotic Disorders
Keywords: Child; Adolescent; Mental Health; Olanzapine; Pharmacokinetics; Pharmacology
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Psychological Well-Being | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
This study will examine the safety and effectiveness of the antipsychotic drug olanzapine in children and adolescents with bipolar disorder or psychosis.

DETAILED DESCRIPTION:
Numerous advancements in mental health treatment have been made over the past decade. Unfortunately, these advancements have focused on adults and have not been fully extended to children and adolescents. With limited pediatric information on the pharmacokinetics and pharmacodynamics for drugs used to treat mental health problems, psychiatrists are prescribing drugs for children using data extrapolated from adults, which may lead to potentially life-threatening results. Olanzapine is widely prescribed to treat both children and adults. This study will determine the safety and effectiveness of olanzapine in children and adolescents with mental health disorders. The study will also compare the effects of gender, development, body composition, and metabolic genotype and phenotype on how olanzapine works.

All participants will receive olanzapine for up to 8 weeks. Blood collection will occur at each weekly study visit. On Visit 1, participants will receive their first dose of olanzapine and repeated blood collection will occur every hour for 24 hours. Blood collection will be used to determine the time it takes for olanzapine to be absorbed into the body, its duration of action, the extent of its distribution in the body, the manner in which it is excreted from the body, and its effects on organs of the body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder with mania, mixed mania, or psychosis not otherwise specified
* Meet certain laboratory result requirements
* Have taken either lithium or valproate for 4 weeks or longer with no or only partial response
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* History of other serious unstable illness requiring medication
* Diabetes mellitus
* Abnormal physical examination and electrocardiogram (EKG) results
* At risk for suicide or homicide (based on an assessment of suicidal history, intent or plan, mental state, mood, and substance use)
* IQ less than 65
* History of organic brain disease or seizure disorder
* Recent exposure to an infectious disease, such as tuberculosis (TB) or meningitis
* Current use of drugs that may interfere with the metabolism of olanzapine and unwilling to discontinue use during the study
* Body mass index (BMI) less than the 5th OR greater than the 95th percentile for age and gender
* History of smoking within 1 year prior to study entry
* Pregnancy or breastfeeding

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68
Dates: Start 2000-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Olanzapine pharmacokinetics, safety, and effectiveness | Measured over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louise G. Cohen, PharmD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Cambridge Health Alliance, Medford, Massachusetts